CLINICAL TRIAL: NCT04966117
Title: A Risk-guided Disease Management and Tele-rehabilitation Program to Reduce Re-admissions in Coronary Artery Disease (Risk-Guided CAD)
Brief Title: Risk-guided Disease Management in Coronary Artery Disease
Acronym: Risk-CAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baker Heart and Diabetes Institute (Other)
Collaborators: Heartwest (Unknown); University of Melbourne (Other); Queen's University, Belfast (Other); Western Health (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 266/21
Record Dates: First submitted 2021-06-29; First posted 2021-07-19 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Coronary Artery Disease; Chronic Disease; Nurse's Role
Keywords: Cardiac rehabilitation; Disease Management Program; Secondary Prevention; Rehospitalization; mHealth
MeSH Terms: conditions — Coronary Artery Disease; Chronic Disease

STUDY DESIGN:
Intervention Model Description: Single site, open, parallel-group randomized controlled trial of a disease management program (intervention group) to reduce hospital readmissions or death compared to usual care (control group)
Who Masked: Outcomes Assessor
Masking Description: There are no other parties who will be masked in the clinical trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Risk-Guided DMP (Experimental): The intervention is a 12 month disease management program after hospital discharge for coronary artery disease that is overseen by a cardiac nurse.
  Interventions: Behavioral: Risk-Guided DMP
- Usual Care (Active Comparator): Usual care patients will receive standard cardiology care.
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Risk-Guided DMP — Patients will be assigned a cardiac nurse to help manage their heart condition who will:
  1. develop a care plan and communicate with the patients' General Practitioner (GP) and cardiologist about management, particularly medications to help control risk factors.
  2. provide health coaching at pre-specified times over 12 months via telehealth (phone or video call) to ensure that patient's take their medications as prescribed and to give health education and guidance on lifestyle changes.
  3. facilitate cardiac rehabilitation via a smart phone or tablet app (called SmartCR). This app monitors health and physical activity, has prompted tasks to do and delivers education via video, audio and written articles. The information from this app can be used by the cardiac nurse during telehealth follow-up.
  4. invite participation to a supervised 6-week group exercise program which will require using our on-site gym.
  Arms: Risk-Guided DMP
Behavioral: Usual Care — Usual care patients will receive standard cardiology care as scheduled that includes adherence to guideline-based care (medications and physical activity), education (self-care), a treatment plan to manage co-morbidities, early post-discharge follow-up/support and routine preventative care.
  Arms: Usual Care

SUMMARY:
Coronary artery disease (CAD) is the number one killer of Australians with a high risk for a recurrent event(s) and hospital readmission. Many of these readmissions can be prevented with better management to control the problem of CAD. A disease management program, led by nurses who interact with other health professionals/providers, can help with education and counselling, taking medications correctly and making healthy lifestyle changes for higher risk patients. Newer models of disease management programs make use of mobile devices (such as an "app") and telehealth (by phone or video call) to monitor and manage health which could facilitate CAD management. Therefore, the aim of this study is to test this type of disease management program (DMP) compared to standard care for reducing hospital readmissions or death in people with CAD who are at high risk of being readmitted. The Investigators envisage that a novel Risk-Guided DMP will be favorable to patients and associated with high-level participation. The Investigators hypothesize that high-risk patients randomized to Risk-Guided CAD will have reduced hospital readmissions or death compared with those randomized to usual care.

DETAILED DESCRIPTION:
The Investigators aim to test a nurse-led, technology-enabled model of health care delivery, called Risk-Guided DMP, to reduce readmissions following CAD, thereby enhancing recovery and survivorship.

The Investigators envisage that a novel Risk-Guided DMP will be favorable to patients and associated with high-level participation. The Investigators hypothesize reduced hospital readmissions or death for high-risk patients randomized to Risk-Guided DMP compared to usual care.

Methods

This proposed study is an effectiveness and feasibility trial of a risk guided DMP to reduce hospital readmissions in CAD patients. The Investigators seek to do this by adopting innovative approaches to:

i) a community-based secondary prevention DMP, ii) supported by a novel m-Health app (SmartCR developed by CardiHab) to address components of a Cardiac Rehabilitation (CR) program, and iii) selection of higher risk patients for appropriate management by validated (PEGASUS-TIMI 54) criteria.

Patients aged 30-74 years who have been hospitalised with CAD will be recruited. Electronic medical records from Western Health (Sunshine or Footscray hospital) will be routinely screened (twice per week) to invite patients to participate. Heartwest cardiologists will also identify patients from their surgical lists.

Baseline measures will include clinical features (including severity and number of affected vessels) and biochemistry (troponin, B-type natriuretic protein, renal function) from medical records; patient self-reported socio-demographic features, cognitive function using the Montreal Cognitive Assessment as an important predictor of readmission, mental health via the Patient Health Questionnaire (PHQ-9) and Generalised Anxiety Disorder (GAD-7) questionnaire and quality of life using the Assessment of Quality of Life (AQoL-8D) questionnaire. Exercise capacity will be quantified by peak oxygen uptake (VO2 peak) and cardiac function will be assessed via two-dimensional echocardiography.

Risk evaluation will be performed by PEGASUS-TIMI 54 criteria for selection of high risk patients [score ≥5] who have an increased risk of a secondary event.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 30 to 74 years; AND
2. Hospitalised with CAD or other eligible cardiac procedure or condition including acute myocardial infarction (STEMI or NSTEMI), unstable angina, coronary artery bypass grafting or percutaneous coronary intervention; AND
3. Defined as higher risk (score >= 5) by PEGASUS-TIMI 54 criteria; AND
4. Eligible for Medicare.

Exclusion Criteria:

1. Inability to provide written informed consent; OR
2. Non-English speaking; OR
3. Inability to attend clinic visits; OR
4. Inability to engage with an app due to low technical literacy or lacking access to a smart phone or wi-fi; OR
5. Hospitalised with a primary diagnosis of heart failure; OR
6. eGFR <30 ml/min/1.73m2 (CKD stage 4 or stage 5); OR
7. Valve disease only; OR
8. Requiring palliative care; OR
9. Concomitant terminal non-cardiac illnesses that could influence 12-month prognosis (e.g. advanced malignancy); OR
10. Participating in another study with a potential but unknown effect on outcome.

Ages: 30 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2021-07-17 (Actual); Primary Completion 2024-10-10 (Actual); Study Completion 2025-07-10 (Actual)

PRIMARY OUTCOMES:
Hospitalization or death | 90 days post discharge
  Unplanned all-cause hospital readmission or death

SECONDARY OUTCOMES:
Hospitalization or death | 30 days post discharge
  Short term unplanned all-cause hospital readmission or death
Provider adherence to best practice guidelines | 12 months post discharge
  Increased prescription of lipid-lowering, anti-hypertensive (e.g. beta-blocker) and antiplatelet agents
Risk factor control - lipids | 12 months post discharge
  Change in LDL-cholesterol (mmol/L)
Risk factor control - blood pressure | 12 months post discharge
  Change in systolic and diastolic blood pressure (mmHg)
Health well-being | 12 months post discharge
  Change in quality of life (via AQoL-8D total scores and 8 dimension scores)

OTHER OUTCOMES:
Mobile Health (mHealth) engagement | 12 months post discharge
  SmartCR (cardiac rehabilitation app) will be evaluated by measures of app engagement by quantifying data entry events and other indicators of program participation/week

CONTACTS AND LOCATIONS:
Overall Officials: Melinda J Carrington, PhD, Principal Investigator — Baker Heart and Diabetes Institute
Locations (1):
- Baker Heart and Diabetes Institute, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Yes
The data to be shared will be all of the individual participant data collected during the trial, after de-identification and underlying published results only. The data will be available to only researchers who provide a methodologically sound proposal, case-by-case basis at the discretion of Principal Investigator. The data will be available for any approved purpose.
Supporting Information: Study Protocol, ICF
Time Frame: Immediately following publication; no end date.
Access Criteria: Access subject to approvals by Principal Investigator.
URL: http://baker.edu.au/research/laboratories/preclinical-disease-prevention

DOCUMENTS (2):
  • Study Protocol (2021-05-19): https://cdn.clinicaltrials.gov/large-docs/17/NCT04966117/Prot_000.pdf
  • Informed Consent Form (2021-05-28): https://cdn.clinicaltrials.gov/large-docs/17/NCT04966117/ICF_001.pdf